CLINICAL TRIAL: NCT00488553
Title: Molecular Epidemiology of Lymphoma Patients
Status: Withdrawn | Type: Observational
Why Stopped: No participants recruited, study discontinued.
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2006-0281
Record Dates: First submitted 2007-06-19; First posted 2007-06-20 (Estimated); Last update posted 2012-02-24 (Estimated); Status verified 2012-02

CONDITIONS: Lymphoma
Keywords: Lymphoma; Epidemiology; Lifestyle Factors; Questionnaire; Survey
MeSH Terms: conditions — Lymphoma | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Subjects will also provide 30 cc of blood. The blood will be genotyped, and the genotype and epidemiological data will be used to evaluate the role of genomic instability (baseline and induced) in the development of lymphomas.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cases: Participants of study with newly diagnosed lymphoma.
  Interventions: Behavioral: Questionnaire
- Control: Participants of study from matched control group.
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — Questions about cancer risk factors, medical history, and family history of cancer.
  Other Names: Survey

SUMMARY:
Primary Objectives:

1. To enroll and obtain, through questionnaires, risk factor information on all study participants to develop detailed demographic, epidemiologic and behavioral profiles.
2. To assess the influence of relevant epidemiologic covariates such as age, gender, smoking and family history of cancer on the panel of susceptibility biomarkers.
3. To evaluate the role of genomic instability in development of lymphomas.

DETAILED DESCRIPTION:
This study will include individuals diagnosed with lymphoma and individuals with no history of cancer. Half of the participants in this study will have lymphoma, and half will have no history of cancer. Information from both groups will be compared to help researchers try to learn which factors may lead to the development of lymphoma.

If you agree to take part in this study, you will be asked to complete a questionnaire at M. D. Anderson. In this questionnaire, you will be asked about your demographics (such as your age, sex, etc.), certain environmental exposures (such as pollution), your medical history, family history, diet, and your past and present smoking and alcohol use habits. This questionnaire should take about 50 minutes to complete.

You will also have about 2 ½ tablespoons of blood drawn for special tests. These tests will look for any biologic factors (such as changes in your DNA) that may be linked to lymphoma. You will not be informed of the results of any of the testing done with your blood samples.

Your participation will be over in this study once your blood has been drawn.

This is an investigational study. Up to 800 participants will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Cases only: Newly diagnosed, previously untreated patients with lymphoma as the primary cancer.
2. Age 18 years and older.
3. Willing to donate 30ml of blood.
4. Willing to complete a self-administered questionnaire.
5. Controls only: No prior cancer.

Exclusion Criteria:

1. Cases only: Prior history of cancer other than lymphoma.
2. Unable to speak or read English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants in this study will include 400 with newly diagnosed lymphoma and 400 matched controls.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2006-08; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
To identify biologic (such as genes) and lifestyle factors that may increase a person's risk of developing lymphoma. | 4 Years

CONTACTS AND LOCATIONS:
Overall Officials: Randa El-Zein, MD, PhD, Principal Investigator — M.D. Anderson Cancer Center

REFERENCES:
- See also: UT MD Anderson Cancer Center Website — http://www.mdanderson.org